CLINICAL TRIAL: NCT05969639
Title: Improving Dietary Habit and Weight Loss in Young Adults With Overweight and Obesity: The Healthy Eating for Young Adults (HEYA) Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National University Health System, Singapore (Other)
Responsible Party: Principal Investigator, Jocelyn Chew, Research Fellow, National University Health System, Singapore
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NUS-IRB-2022-650
Record Dates: First submitted 2023-07-23; First posted 2023-08-01 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The HEYA program is a 12-week app-delivered psychoeducational program that comprises of nutrition education, skills training on self-regulation, and weekly feedback.
  Interventions: Behavioral: HEYA
- Control (No Intervention)

INTERVENTIONS:
Behavioral: HEYA — The HEYA program is a 12-week app-delivered psychoeducational program that comprises of nutrition education, skills training on self-regulation, and weekly feedback.
  Arms: Intervention

SUMMARY:
This study aims to examining the effectiveness of a psychoeducational program (Healthy Eating in Young Adults; HEYA) on improving the dietary habits and body composition (e.g. weight and percentage fat mass) in young adults in Singapore.

ELIGIBILITY:
Inclusion Criteria:

1. have a body mass index (BMI) ≥23kg/m2; and
2. are between the ages of 21 and 35 years old; and
3. can understand and read the English language; and
4. use a smartphone that can download apps; and
5. willing to travel to the National University Singapore.

Exclusion Criteria:

1. Pregnant or lactating; and
2. Participating in a structured weight loss program; and
3. Planning or receiving pharmacotherapy or bariatric surgery within the next 6 months; and
4. Has existing diagnosed mental disorder besides eating disorders.

Ages: 21 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-07-25 (Estimated); Primary Completion 2024-07-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
weight | 0,12,24

CONTACTS AND LOCATIONS:
Locations (1):
- National University of Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No